CLINICAL TRIAL: NCT05907187
Title: Intervention to Promote Cervical Cancer Prevention and Early Detection, and Understand the Role of Plants in HPV. (Research in Ethno-Medicine and Education)
Brief Title: Research in Ethno-Medicine and Education (REMED)
Acronym: REMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Cigna Foundation (Unknown)
Responsible Party: Principal Investigator, Erin Kobetz-Kerman, PhD, MPH, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20170445; NCI-2023-00177 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cervical Cancer; Human Papilloma Virus; HPV; Human Papillomavirus Infection
Keywords: Twalet Deba
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Twalet Deba Group (Experimental): Participants will receive cervical cancer prevention education, and provide self-administered vaginal or cervical specimens and provide specimens of plants, plant-products or herbs most commonly used in the intravaginal cleansing practice of twalet deba. Total expected participation is about 30 days.
  Interventions: Behavioral: Cervical Cancer Prevention Education

INTERVENTIONS:
Behavioral: Cervical Cancer Prevention Education — Participants will receive in-person, one-time health education on the importance of cervical cancer screening using a short intervention/educational script; and motivation to encourage women to have human papillomavirus (HPV) screening. Participants will also be informed of the nature and risks of HPV infection, and the importance of seeing a doctor including having a gynecologic exam.

SUMMARY:
The purpose of this study is to gain information about intravaginal practices, like intravaginal "twalet deba", among Haitian women living in South Florida. Intravaginal "twalet deba" may include douching, cleaning inside the vagina with different kinds of products, or using steam/vapor that enter the vagina. The investigators want to help learn the best way to increase early detection and/or prevention for cervical cancer. The investigators would like to know what plants, herbs, commercial products and medicines are used in these practices, how these products are prepared, applied, why these products are used, and how these products affect the vagina and cervix.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Self-identifies as Haitian or Haitian-American
* Resident of Miami-Dade, Broward or Palm Beach County
* Currently engages in regular intravaginal cleansing practices that involve more than just water alone
* No history of hysterectomy
* Speaks Creole or English

Exclusion Criteria:

* Are adults unwilling or unable to provide consent
* Individuals less than 18 years of age
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Plant products used for intravaginal twalet deba. | Up to 30 days
  Identification of the most commonly used plant products for intravaginal twalet deba as measured by the Research in Ethno-Medicine and Education (REMED) tool.
Methods of using plant products for intravaginal twalet deba. | Up to 30 days
  Identification of the most commonly used methods of using plant products for intravaginal twalet deba as measured by the Research in Ethno-Medicine and Education (REMED) tool.
Cultural beliefs surrounding the practice of intravaginal twalet deba. | Up to 30 days
  Identification of the most commonly held cultural beliefs surrounding the practice of intravaginal twalet deba as measured by the Research in Ethno-Medicine and Education (REMED) tool.
Health access for cervical cancer screening as measured by REMED tool | Up to 30 days
  The REMED tool will collect information regarding early detection and prevention of cervical cancer among underserved communities.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Kobetz-Kerman, PhD, MPH, Principal Investigator — University of Miami
Locations (1):
- Martine Poitevien, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No